CLINICAL TRIAL: NCT03155451
Title: Plasma ctDNA Detection in Diagnosis of Epithelial Ovarian Cancer.
Acronym: ctDNA_EOC
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wang Yu, M.D., RenJi Hospital
Other Study IDs: [2017]012
Record Dates: First submitted 2017-05-13; First posted 2017-05-16 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epithelial ovarian cancer: patients receive the ctDNA methylation markers screening
  Interventions: Diagnostic Test: methylation markers screening

INTERVENTIONS:
Diagnostic Test: methylation markers screening — ctDNA extraction from plasma samples;bisulfite-treated DNA;DNA methylation levels by deep sequencing-Sequencing; data analysis

SUMMARY:
Epithelial ovarian cancer constitutes one of the most common gynecological malignancies.Because the ovaries lie in the deep pelvic cavity,most ovarian cancer patients are asymptomatic, rendering the majority often diagnosed at an advanced stage.ctDNA in cancer patients often bears similar genetic and epigenetic features to the related tumor DNA.This study aims to detect plasma ctDNA in Diagnosis of Epithelial Ovarian Cancer.

DETAILED DESCRIPTION:
Epithelial ovarian cancer constitutes one of the most common gynecological malignancies, with an incidence rate of 3-12/100 000 woman per year. Because the ovaries lie in the deep pelvic cavity,most ovarian cancer patients are asymptomatic, rendering the majority often diagnosed at an advanced stage. Liquid biopsy, which is meant to detect cancers by sequencing the DNA in a few drops of a person's blood. It may detect cancers early, even before symptoms arise, when there is just a few cells in the blood circulation.

ctDNA in cancer patients often bears similar genetic and epigenetic features to the related tumor DNA. There is evidence that some of the ctDNA originates from tumor tissue. This, and the fact that ctDNA can easily be isolated from the circulation and other body fluids of patients, makes it a promising candidate as a non-invasive biomarker of cancer.

This study aims to detect plasma ctDNA in Diagnosis of Epithelial Ovarian Cancer.

ELIGIBILITY:
Inclusion Criteria:

* people aged 18years to 80years;
* Diagnosis of ovarian cancer is confirmed by two Pathologists independently;
* Pregnancy tests are negative.

Exclusion Criteria:

* With other type of malignancies;
* someone who refuse to participate the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women
Study Population: consecutive colletion of patinets with ovarian cancer treatment at our clinical centre
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Pathological diagnosis of ovarian lumps | One week after surgery
  Pathological diagnosis of ovarian lumps，including immunohistochemical information and HE staining information.

SECONDARY OUTCOMES:
sensitivity (true positive rate) | 2 year
  The proportion of persons with disease who have a positive test (positive test results among persons with disease)
Specificity (true negative rate) | 2 year
  The proportion of persons without disease who have a negative test (negative test results among persons without disease)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wang, M.D., Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wen L, Li J, Guo H, Liu X, Zheng S, Zhang D, Zhu W, Qu J, Guo L, Du D, Jin X, Zhang Y, Gao Y, Shen J, Ge H, Tang F, Huang Y, Peng J. Genome-scale detection of hypermethylated CpG islands in circulating cell-free DNA of hepatocellular carcinoma patients. Cell Res. 2015 Nov;25(11):1250-64. doi: 10.1038/cr.2015.126. Epub 2015 Oct 30. PMID 26516143
- [Background] Nick AM, Coleman RL, Ramirez PT, Sood AK. A framework for a personalized surgical approach to ovarian cancer. Nat Rev Clin Oncol. 2015 Apr;12(4):239-45. doi: 10.1038/nrclinonc.2015.26. Epub 2015 Feb 24. PMID 25707631